CLINICAL TRIAL: NCT04338802
Title: Efficacy and Safety of Nintedanib Ethanesulfonate Soft Capsule in the Treatment of Pulmonary Fibrosis in Patients With Moderate to Severe COVID-9(COVID 19) : a Single-center, Randomized, Placebo-controlled Study
Brief Title: Efficacy and Safety of Nintedanib in the Treatment of Pulmonary Fibrosis in Patients With Moderate to Severe COVID -19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huilan Zhang (Other)
Responsible Party: Sponsor-Investigator, Huilan Zhang, Director of Respiratory and Critical Care Medicine , Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: huilanz Zhang
Record Dates: First submitted 2020-04-01; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; Nintedanib; Safety; Effect of Drugs
MeSH Terms: conditions — COVID-19 | interventions — nintedanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Empty capsules with the same appearance and ingredients as Nintedanib soft capsules: one capsule at a time, twice a day, with an interval of about 12 hours each time. Continuous medication for 8 weeks.
  Interventions: Other: Placebo
- Nintedanib group (Experimental): Nintedanib cloth sulfonate soft capsule treatment: According to the drug manual recommendation, give Nintedanib cloth sulfonate soft capsule 150mg twice daily with an interval of about 12 hours each time. Continuous medication for 8 weeks.
  Interventions: Drug: Nintedanib 150 MG

INTERVENTIONS:
Drug: Nintedanib 150 MG — Nintedanib cloth sulfonate 150 mg, twice a day, about 12 hours apart. Continuous medication for 8 weeks.
  Arms: Nintedanib group
Other: Placebo — Empty capsules with the same appearance and ingredients as Nidanib soft capsules: one capsule at a time, twice a day, with an interval of about 12 hours each time. Continuous medication for 8 weeks.
  Arms: Placebo group

SUMMARY:
This center intends to conduct a single-center, randomized, placebo-controlled study to evaluate the effectiveness and safety of Nintedanib ethanesulfonate soft capsule in the treatment of pulmonary fibrosis in patients with moderate to severe COVID-19.

DETAILED DESCRIPTION:
This center intends to conduct a single-center, randomized, placebo-controlled study to evaluate the effectiveness and safety of Nintedanib ethanesulfonate soft capsule in the treatment of pulmonary fibrosis in patients with moderate to severe COVID-19. The number of cases is estimated based on the following:

This exploratory trial is expected to complete 80 case studies (randomly divided into control group and test group each with 40 cases), and the expected drop-out rate is not more than 20%, so the total number of cases is 96. Placebo control group:

Empty capsules with the same appearance and ingredients as Nintedanib soft capsules: one capsule at a time, twice a day, with an interval of about 12 hours each time. Continuous medication for 8 weeks.

Nintedanib Nintedanib cloth sulfonate soft capsule treatment: According to the drug manual recommendation, give Nintedanib cloth sulfonate soft capsule 150mg twice daily with an interval of about 12 hours each time, with food. Continuous medication for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old (including 18 and 70 years old), regardless of gender;
2. Infection with new coronavirus pneumonia was confirmed by throat swab nucleic acid test. Patients with severe and critical illness were clinically judged. The symptoms of acute infection have been alleviated after treatment (at least 14 days after onset, no fever for more than 3 days), and the disease is recovering Within three months;
3. CT examination of patients with multiple fibrotic shadows in both lungs;
4. Blood routine, liver, and kidney functions are within the controllable range: such as the normal upper limit of plasma total bilirubin and creatinine ≤ 1.5 times; AST, ALT, LDH ≤ 2 times the normal upper limit; sufficient hematopoietic function: such as white blood cells ≥4.0 × 109 / L, platelets ≥100 × 109 / L;
5. Signed informed consent.

Exclusion Criteria:

1. Previous history of chronic bronchitis, emphysema, interstitial lung disease or pulmonary heart disease;
2. Combining with other serious diseases: such as those who have suffered myocardial infarction and uncontrollable diabetes within 6 months, and are considered unsuitable to participate in the trial;
3. People with active peptic ulcer;
4. Patients during pregnancy and lactation
5. Patients with mental illness or others who cannot cooperate effectively;
6. Researcher judges uncomfortable to participate in trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-04-02 (Estimated); Primary Completion 2020-05-04 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in forced vital capacity (FVC) | 8 weeks
  Changes in forced vital capacity (FVC) after treatment compared to baseline.

SECONDARY OUTCOMES:
Changes in carbon monoxide dispersion (DLco%) | 8 weeks
  Changes incarbon monoxide dispersion (DLco%) after treatment compared to baseline.
Changes in the six-minute walk test (6MWT) | 8 weeks
  Changes in the six-minute walk test (6MWT) after treatment compared to baseline.
Changes in High resolution CT score | 8 weeks
  Changes in High resolution CT score after treatment compared to baseline.The minimum and maximum values are 0 and 25 , and higher scores mean a worse outcome. As for the score, it is the expected value and will be determined according to the actual result

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flaherty KR, Wells AU, Cottin V, Devaraj A, Walsh SLF, Inoue Y, Richeldi L, Kolb M, Tetzlaff K, Stowasser S, Coeck C, Clerisme-Beaty E, Rosenstock B, Quaresma M, Haeufel T, Goeldner RG, Schlenker-Herceg R, Brown KK; INBUILD Trial Investigators. Nintedanib in Progressive Fibrosing Interstitial Lung Diseases. N Engl J Med. 2019 Oct 31;381(18):1718-1727. doi: 10.1056/NEJMoa1908681. Epub 2019 Sep 29. PMID 31566307
- [Background] Richeldi L, du Bois RM, Raghu G, Azuma A, Brown KK, Costabel U, Cottin V, Flaherty KR, Hansell DM, Inoue Y, Kim DS, Kolb M, Nicholson AG, Noble PW, Selman M, Taniguchi H, Brun M, Le Maulf F, Girard M, Stowasser S, Schlenker-Herceg R, Disse B, Collard HR; INPULSIS Trial Investigators. Efficacy and safety of nintedanib in idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2071-82. doi: 10.1056/NEJMoa1402584. Epub 2014 May 18. PMID 24836310
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Xie L, Liu Y, Fan B, Xiao Y, Tian Q, Chen L, Zhao H, Chen W. Dynamic changes of serum SARS-coronavirus IgG, pulmonary function and radiography in patients recovering from SARS after hospital discharge. Respir Res. 2005 Jan 8;6(1):5. doi: 10.1186/1465-9921-6-5. PMID 15638943